CLINICAL TRIAL: NCT05640011
Title: Clinical Validation of an Artificial Intelligence Algorithm to Help Interpret Mammograms
Acronym: ALGO-MAMMO
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7964
Record Dates: First submitted 2022-11-25; First posted 2022-12-07 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2022-11

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Mammography; Artificial intelligence; Tumor detection on mammograms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This aims to clinically validate, on a large population, a tumor detection aid software which has already been trained on a representative French population (from several hospital centers and liberals from several departments in the west and east of France).

This population consists of 1000 patients who have been treated for breast cancer (histologically proven by breast biopsy) and whose investigators have mammograms performed at the time of diagnosis. The control population consists of the unaffected breast of each patient (with the exception of the rare cases of bilateral cancers).

This innovative software has the main feature of recognizing healthy breast tissue, allowing the radiologist to focus on breast tissue at risk, improving the management of medical time and the management of "difficult" files.

ELIGIBILITY:
Inclusion Criteria:

* Adult woman (40 to 75 years old)
* Treatment at the University Hospitals of Strasbourg between 2010 and 2020 for breast cancer
* including mammography and histological evidence available
* Patient who has already given her consent for the reuse of her anonymous data for research purposes

Exclusion Criteria:

* Woman who expressed her opposition to participating in the study

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult woman (40 to 75 years old) treated at the University Hospitals of Strasbourg between 2010 and 2020 for breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
Evaluate the diagnostic performance (sensitivity, specificity) for operator tumor detection assisted by mammographic diagnostic aid software, and compare it to the diagnostic performance of an unassisted operator. | Files analysed retrospectively from January 01, 2010 to January 01, 2020 will be examined
  This assessment is based on contouring the tumor area on mammograms.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Radiologie 1 - CHU de Strasbourg - France, Strasbourg, France